CLINICAL TRIAL: NCT00546962
Title: Tissue Bank for Pulmonary Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Thomas Martin, MD, Childrens Hospital Boston
Other Study IDs: 05-02-014R
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this research study is to collect and store the specimens that are left over after patients undergo tests ordered by their physicians. These specimens will be used at a later time by researchers in the Pulmonary Division to develop a better understanding of pulmonary diseases or for the development of new treatments. Typical research studies that will be conducted on the stored tissue, fluid, or bacteria from the patient sample involve obtaining bacterial cultures, measurement of inflammatory markers, and examination of the characteristics of the tissue. Other similar tests may be done in the future; however, these tests have not all been determined at this time. It is important to note that no genetic testing will be performed on any samples that are obtained as part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Open

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic Fibrosis Patients, Pulmonary Patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States